CLINICAL TRIAL: NCT05200858
Title: Transcutaneous Electrical Nerve Stimulation For Lower Extremity In Patients With Neurogenic Pain - A Proof Of Concept Randomized Clinical Trial
Brief Title: Transcutaneous Electrical Nerve Stimulation (TENS) in Patients With Postacute Sequelae of Sars-CoV-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: NeuroMetrix, Inc. (Industry)
Responsible Party: Principal Investigator, Bijan Najafi, PhD, Professor of Surgery, Baylor College of Medicine
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: H-50753-A
Record Dates: First submitted 2021-12-28; First posted 2022-01-21 (Actual); Results first posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Postacute Sequelae of Sars-CoV-2; Post-Acute COVID-19 Syndrome; Widespread Chronic Pain; Fatigue Syndrome, Chronic; Gait, Unsteady
Keywords: Transcutaneous nerve electrical stimulation; Pain; Fatigue
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Chronic Pain; Fatigue Syndrome, Chronic; Gait Disorders, Neurologic; Pain; Fatigue | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Participants, who satisfy the inclusion and exclusion criteria and sign the informed consent form will be randomly assigned with ratio of 1:1 into two groups. One group will utilize TENS high-dose devices (Intervention group, IG); the other group will utilize TENS low-dose devices (Placebo group, PG).
  Both groups will receive their respective devices at the initial visit (BL) and will be asked to return in 4 weeks for follow-up assessment (4W visit). At this 4 week visit, study participants will be unblinded and the IG will keep their high-dose device, while the PG will switch from low-dose to high-dose TENS device. Study participants will return for a final in-person visit at the 8th week (8W), which will include the assessments described above. Throughout this 8-week period the participants may receive follow-up phone calls assessing their compliance. All subjects will keep the commercial (high-dose TENS) device after completion of the 8-week study.
Who Masked: Participant, Care Provider
Masking Description: Devices may be high-dose (delivering 100% of the dose) or low-dose (delivering 10% of the dose) TENS
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Intervention Group at 4 weeks (blinded phase) (Active Comparator): The IG will be undergoing Transcutaneous Electrical Nerve Stimulation (TENS) therapy with a functional device during a blinded period of 4 weeks.
  The functional device elicits 1 hour of TENS per session. Each session lasts 1 hour (100% of dose). To deliver TENS, a band strap with hydrogel pads will be placed around the calf muscle of one lower-extremity alternating to the other side in a weekly basis.
  Interventions: Device: TENS - high-dose
- Placebo Group at 4 weeks (blinded phase) (Placebo Comparator): The PG will be undergoing Transcutaneous Electrical Nerve Stimulation (TENS) therapy with a placebo device during a blinded period of 4 weeks. The placebo device is identical to the functional device in all respects except that it delivers 6 minutes of TENS therapy per session (10% out of 60 minutes).
  Interventions: Device: TENS - low-dose
- Intervention Group at 8 weeks (unblinded phase) (Active Comparator): After 4 weeks, the IG will be unblinded, and will continue to receive high-dose TENS with a functional device for additional 4 weeks until completing 8 weeks.
  The functional device elicits 1 hour of TENS per session. Each session lasts 1 hour (100% of dose). To deliver TENS, a band strap with hydrogel pads will be placed around the calf muscle of one lower-extremity alternating to the other side in a weekly basis.
  Interventions: Device: TENS - high-dose
- Placebo Group at 8 weeks (unblinded phase) (Active Comparator): After 4 weeks, the PG will be unblinded and will switch to a high-dose TENS with a functional device for additional 4 weeks until completing 8 weeks.
  The functional device elicits 1 hour of TENS per session. Each session lasts 1 hour (100% of dose). To deliver TENS, a band strap with hydrogel pads will be placed around the calf muscle of one lower-extremity alternating to the other side in a weekly basis.
  Interventions: Device: TENS - high-dose

INTERVENTIONS:
Device: TENS - high-dose — Subjects will receive a functional TENS device (delivers 100% of the dose) to wear for 3-5 hours per day.
  Other Names: functional; commercial
  Arms: Intervention Group at 4 weeks (blinded phase); Intervention Group at 8 weeks (unblinded phase); Placebo Group at 8 weeks (unblinded phase)
Device: TENS - low-dose — Subjects will receive a placebo TENS device (delivers 10% of the dose) to wear for 3-5 hours per day.
  Other Names: placebo; sham
  Arms: Placebo Group at 4 weeks (blinded phase)

SUMMARY:
The purpose of the pilot study is to examine acceptability and proof of concept effectiveness of a wireless TENS technology to address PASC associated FM. Sample size (n=30) is convenient and designed to explore acceptability and feasibility. Participants, who satisfy the inclusion and exclusion criteria and sign the informed consent form will be randomly assigned with ratio of 1:1 into two groups. One group will utilize TENS high-dose devices (Intervention group, IG); the other group will utilize TENS low-dose devices (Placebo group, PG). The baseline measurements will be performed, and the patients will take the programmed device home for a duration of 4 weeks. Then, the patients will come back after four weeks (4W). At this 4th week visit, both groups will be unblinded and the IG will keep their high-dose TENS device and the PG group will switch from a low-dose TENS to a high-dose TENS device. Both groups will continue to deliver 3-5 hour of stimulation daily, until their final 8th week follow up visit (8W). The primary outcome will be pain. Secondary outcomes include fatigue, limb strength and perfusion, gait assessment (cadence, stride time, double support), balance, pulse oximetry, and quality of life. The coordinator will utilize a weekly spreadsheet showing utilization (therapy sessions/day, logged in the Quell health Cloud) so compliance can be monitored and those that are not using the device can be encouraged.

DETAILED DESCRIPTION:
Postacute Sequelae of Sars-CoV-2 (PASC) is an emerging entity that has been clearly recognized by musculoskeletal pain, fatigue, cognitive, and sleep disturbances, among other symptoms, in patients who have recovered from severe Sars-CoV-2 infection. Hospitalized survivors have reported a significant excess burden of many of these symptoms up to 8 months after discharge. Particularly in the lower extremity, musculoskeletal illness has been associated with prolonged immobilization, high-risk comorbidities, and the use of glucocorticoids that is commonly administered to these patients. These manifestations are the cardinal symptoms of fibromyalgia (FM), a condition thought to be caused by hyperactive sensory signaling due to central sensitization as well as deficient endogenous pain inhibition, triggered among others, by viral infections. Consequently, FM sequelae are one of the most common long-term complications seen in PASC. Thus, it is expected to impose a serious burden on different medical specialties in a near future. In a population that has persistent lack of symptom resolution such as FM, adherence to therapy could be challenging. Patients with constant pain, fatigue, and sleep disturbances, are difficult to keep motivated, especially those pain-medication dependents that often present low quality of life. One practical solution to address the symptomatology characteristic of FM is the use of transcutaneous electrical stimulation therapy (TENS). Studies have demonstrated its ability to manage pain and fatigue in patients with peripheral neuropathy and FM, and has shown to effectively improve lower-extremity perfusion and oxygen delivery in patients with ischemic lesions. However, TENS has not yet been explored for PASC. Since this technology is dose-dependent, the investigators propose a practical daily-basis therapy that patients with persistent associated FM due to previous COVID-19 infection could apply at home, thus, addressing PASC without relying only on medication. In this matter, Neurometrix Inc. (Woburn, MA, USA) has created a wireless TENS device (Quell®) to address pain, gait, sleep, and fatigue. This technology is placed in the lower-extremity and works through the stimulation of nerves that carry non-painful sensations (A-beta fibers) by closing a neurological "gate" in the spinal cord, thus, reducing transmission from pain nerves (A-delta and C fibers) to the brain. This device utilizes a wireless technology manageable through a smart phone application (Quell App) that also tracks symptom-status. Moreover, Baylor College of Medicine has created the Post-COVID-19 Clinic (McNair Campus, BCM St Luke's, Houston, TX, USA) supervised by specialists in critical and pulmonary care. This Clinic has a high volume of patients that present with PASC, particularly those with associated FM (i.e., persistent muscle pain, fatigue, weakness, atrophy, sleep problems, and/or anxiety). Therefore, the investigators believe Baylor institution is a suitable place to perform this pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Previous COVID-19 infection
* Persistent symptoms of pain, fatigue, weakness, or poor gait and balance that were not present before COVID-19 infection
* Willing to attend clinic for assessments

Exclusion Criteria:

* Severe cognitive decline reduces their ability to interact with the TENS mobile app
* Major visual or hearing weakness reduces the ability to interact with TENS mobile app
* Unable to walk independently for a distance of 10 meter
* Major foot problems such as active lower extremity wounds, major foot deformity (e.g., Charcot Foot), previous major amputations, and claudication
* Demand-type cardiac pacemaker, implanted defibrillator, or other implanted electronic devices; and any conditions that may interfere with outcomes or increase the risk of the use TENS based on the judgement of clinicians

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Group (AG) Blinded Phase: The IG will be undergoing Transcutaneous Electrical Nerve Stimulation (TENS) therapy with a functional device during 4 weeks.
  The functional device elicits 1 hour of TENS per session. Each session lasts 1 hour (100% of dose). To deliver TENS, a band strap with hydrogel pads will be placed around the calf muscle of one lower-extremity alternating to the other side in a weekly basis.
- Placebo Group (PG) Blinded Phase: The PG will be undergoing Transcutaneous Electrical Nerve Stimulation (TENS) therapy with a placebo device during 4 weeks. The placebo device is identical to the functional device in all respects except that it delivers 6 minutes of TENS therapy per session (10% out of 60 minutes).
- Active Group (AG) Unblinded Phase: After 4 weeks, the IG will be unblinded, and will continue to receive high-dose TENS with a functional device for additional 4 weeks until completing 8 weeks.
  The functional device elicits 1 hour of TENS per session. Each session lasts 1 hour (100% of dose). To deliver TENS, a band strap with hydrogel pads will be placed around the calf muscle of one lower-extremity alternating to the other side in a weekly basis.
- Placebo Group (PG) Unblinded Phase: After 4 weeks, the PG will be unblinded and will switch to a high-dose TENS with a functional device for additional 4 weeks until completing 8 weeks.
  The functional device elicits 1 hour of TENS per session. Each session lasts 1 hour (100% of dose). To deliver TENS, a band strap with hydrogel pads will be placed around the calf muscle of one lower-extremity alternating to the other side in a weekly basis.
Period: Blinded Phase (4 Weeks)
Arm/Group | Active Group (AG) Blinded Phase | Placebo Group (PG) Blinded Phase | Active Group (AG) Unblinded Phase | Placebo Group (PG) Unblinded Phase
Started | 15 | 15 | 0 | 0
Completed | 12 | 13 | 0 | 0
Not Completed | 3 | 2 | 0 | 0
Not completed — Lost to Follow-up | 3 | 2 | 0 | 0
Period: Unblinded Phase (4 Weeks)
Arm/Group | Active Group (AG) Blinded Phase | Placebo Group (PG) Blinded Phase | Active Group (AG) Unblinded Phase | Placebo Group (PG) Unblinded Phase
Started | 0 (All patients were unblinded at the end of the first 4 weeks and all were given the active device to use in the last 4 weeks (unblinded phase).) | 0 (No patients were using the placebo device in the final 4 weeks of the study.) | 12 | 13
Completed | 0 | 0 | 10 | 10
Not Completed | 0 | 0 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Placebo Group (PG): Placebo Group (PG) The PG (n=15) will be undergoing TENS therapy with a sham device as described in the AG. The sham device is identical to the active device in all respects except that it stimulates for 6 minutes during each therapy session instead of 60 minutes, and is therefore 10% of the dose.
  Electrical Stimulation - Placebo: Subjects will receive a placebo electrical stimulation device (delivers 10% of the dose) to wear for 1 hour daily for up to 4 weeks.
- Active Group (AG): Active group (AG). The AG (n=15) will be undergoing TENS therapy with an active device during 4 weeks. To deliver TENS, a band strap with hydrogel pads will be placed around the calf muscle of one lower-extremity alternating to the other side in a weekly basis.
  Electrical Stimulation - Active: Subjects will receive an active electrical stimulation device (delivers 100% of the dose) to wear for 1 hour daily for up to 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo Group (PG) | Active Group (AG) | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.38 (11.79) | 51.08 (12.32) | 45.28 (12.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 4 | 2 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 1 | 2 | 3
  Hispanic | 2 | 3 | 5
  Asian | 2 | 0 | 2
  White | 6 | 6 | 12
  Unknown | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 25
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.76 (5.98) | 27.72 (7.92) | 27.74 (6.95)
High Blood Pressure [Count of Participants; unit: Participants] | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Functional Interference From Pain From Baseline to 4 Weeks (Blinded Phase)
Description: Pain will be assessed with a validated questionnaire called Brief Pain Inventory interference composite score (BPI-I). The maximum score is 10, meaning pain completely interferes, while the minimum score is zero, meaning pain does not interfere.
Time Frame: baseline to 4 weeks
Population: Blinded phase of the study at 4 weeks.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Intervention Group: The IG will be undergoing Transcutaneous Electrical Nerve Stimulation (TENS) therapy with a functional device during 4 weeks.
  The functional device elicits 1 hour of TENS per session. Each session lasts 1 hour (100% of dose). To deliver TENS, a band strap with hydrogel pads will be placed around the calf muscle of one lower-extremity alternating to the other side in a weekly basis.
  TENS - Functional: Subjects will receive a functional TENS device (delivers 100% of the dose) to wear for 1 hour daily for up to 4 weeks.
- Placebo Group: The PG will be undergoing Transcutaneous Electrical Nerve Stimulation (TENS) therapy with a placebo device during 4 weeks. The placebo device is identical to the functional device in all respects except that it delivers 6 minutes of TENS therapy per session (10% out of 60 minutes).
  TENS - Placebo: Subjects will receive a placebo TENS device (delivers 10% of the dose) to wear for 1 hour daily for up to 4 weeks.
Arm/Group | Intervention Group | Placebo Group
Number analyzed (Participants) | 11 | 12
score on a scale | 0.454 (0.503) | 0.198 (0.503)

2. Secondary Outcome: Mean Change in Pain Severity From Baseline to 4 Weeks (Blinded Phase)
Description: Pain severity will be assessed using the Brief Pain Inventory questionnaire composite score for severity. The maximum score is 10, meaning pain as bad as one can imagine, while the minimum score is zero, meaning no pain.
Time Frame: Baseline to 4 weeks
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Intervention Group at 4 Weeks (Blinded Phase): The IG will be undergoing Transcutaneous Electrical Nerve Stimulation (TENS) therapy with a functional device during a blinded period of 4 weeks.
  The functional device elicits 1 hour of TENS per session. Each session lasts 1 hour (100% of dose). To deliver TENS, a band strap with hydrogel pads will be placed around the calf muscle of one lower-extremity alternating to the other side in a weekly basis.
  TENS - high-dose: Subjects will receive a functional TENS device (delivers 100% of the dose) to wear for 3-5 hours per day.
Arm/Group | Intervention Group at 4 Weeks (Blinded Phase) | Placebo Group at 4 Weeks (Blinded Phase)
Number analyzed (Participants) | 10 | 11
score on a scale | 1.184 (0.815) | 0.289 (0.255)

3. Secondary Outcome: Mean Change in Functional Interference From Fatigue From Baseline to 4 Weeks (Blinded Phase)
Description: Functional interference from fatigue will be assessed calculating the Global Fatigue Index (GFI) obtained from a validated questionnaire called Multidimensional Assessment Fatigue, which has a minimum score of 0 (no fatigue) and a maximum sore of 100 (severe fatigue).
Time Frame: Baseline to 4 weeks
Population: Blinded phase of the study.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Active Group (AG): The IG will be undergoing Transcutaneous Electrical Nerve Stimulation (TENS) therapy with a functional device during 4 weeks.
  The functional device elicits 1 hour of TENS per session. Each session lasts 1 hour (100% of dose). To deliver TENS, a band strap with hydrogel pads will be placed around the calf muscle of one lower-extremity alternating to the other side in a weekly basis.
- Placebo Group (PG): The PG will be undergoing Transcutaneous Electrical Nerve Stimulation (TENS) therapy with a placebo device during 4 weeks. The placebo device is identical to the functional device in all respects except that it delivers 6 minutes of TENS therapy per session (10% out of 60 minutes).
Arm/Group | Active Group (AG) | Placebo Group (PG)
Number analyzed (Participants) | 11 | 10
score on a scale | 2.821 (1.504) | 2.231 (3.207)

4. Secondary Outcome: Stride Time at 4 Weeks During a Simple Walking Task (Blinded Phase)
Description: Stride time will be measured with wearable sensors (LEGSys, BioSensics, MA) during a free walking task (single task) using normal pace for 30 ft. Stride time is defined as the period elapsed between the first contact of two consecutive footsteps of the same foot expressed in seconds.
Time Frame: at 4 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Active Group (AG) | Placebo Group (PG)
Number analyzed (Participants) | 9 | 12
seconds | 1.13 (0.03) | 1.16 (0.03)

5. Secondary Outcome: Cadence at 4 Weeks During a Simple Walking Task (Blinded Phase)
Description: Cadence will be measured with wearable sensors (LEGSys, BioSensics, MA) during a free walking task (single task) using normal pace for 30 ft. Cadence is defined as rate of number of steps per minute.
Time Frame: at 4 weeks
Population: blinded phase
Measure: Mean (Standard Deviation); unit: steps/min
Arm/Group | Active Group (AG) | Placebo Group (PG)
Number analyzed (Participants) | 11 | 12
steps/min | 106.42 (10.35) | 105.90 (10.13)

6. Secondary Outcome: Double Support Phase at 4 Weeks During a Simple Walking Task (Blinded Phase)
Description: Double Support Phase will be measured with wearable sensors (LEGSys, BioSensics, MA) during a free walking task (single task) using normal pace for 30 ft. Double support phase is defined as percentage time when both feet are simultaneously in contact with the ground during a single stride.
Time Frame: at 4 weeks
Population: blinded phase
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Active Group (AG) | Placebo Group (PG)
Number analyzed (Participants) | 11 | 12
percentage of time | 22.84 (3.98) | 22.64 (4.08)

7. Secondary Outcome: Cadence at 4 Weeks During a Dual Walking Task (Blinded Phase)
Description: Cadence will be measured with wearable sensors (LEGSys, BioSensics, MA) during a dual walking task (participants asked to count backwards by two while walking) using normal pace for 30 ft. Cadence is defined as rate of number of steps per minute.
Time Frame: at 4 weeks
Population: blinded phase
Measure: Mean (Standard Deviation); unit: steps/min
Arm/Group | Active Group (AG) | Placebo Group (PG)
Number analyzed (Participants) | 10 | 12
steps/min | 103.40 (17.36) | 103.40 (14.84)

8. Secondary Outcome: Cadence at 4 Weeks During a Fast Walking Task (Blinded Phase)
Description: Cadence will be measured with wearable sensors (LEGSys, BioSensics, MA) during a fast walking task (participants asked to walk at a slightly faster pace) for 30 ft. Cadence is defined as rate of number of steps per minute.
Time Frame: at 4 weeks
Population: blinded phase
Measure: Mean (Standard Deviation); unit: steps/min
Arm/Group | Active Group (AG) | Placebo Group (PG)
Number analyzed (Participants) | 11 | 11
steps/min | 122.57 (15.87) | 122.57 (14.80)

9. Other Pre Specified Outcome: Stride Time at 4 Weeks During a Dual Walking Task (Blinded Phase)
Description: Stride time will be measured with wearable sensors (LEGSys, BioSensics, MA) during a dual walking task (participants asked to count backwards by two while walking) using normal pace for 30 ft. Stride time is defined as the period elapsed between the first contact of two consecutive footsteps of the same foot expressed in seconds.
Time Frame: at 4 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Intervention Group at 4 Weeks (Blinded Phase) | Placebo Group at 4 Weeks (Blinded Phase)
Number analyzed (Participants) | 10 | 12
seconds | 1.19 (0.21) | 1.19 (0.20)

10. Other Pre Specified Outcome: Stride Time at 4 Weeks During a Fast Walking Task (Blinded Phase)
Description: Stride time will be measured with wearable sensors (LEGSys, BioSensics, MA) during a fast walking task (participants asked to walk at a slightly faster pace) for 30 ft. Stride time is defined as the period elapsed between the first contact of two consecutive footsteps of the same foot expressed in seconds.
Time Frame: at 4 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Intervention Group at 4 Weeks (Blinded Phase) | Placebo Group at 4 Weeks (Blinded Phase)
Number analyzed (Participants) | 11 | 11
seconds | 1.00 (0.13) | 1.00 (0.12)

11. Other Pre Specified Outcome: Gastrocnemius Muscle Endurance (Muscle Sustained Contraction) in Response to Electrical Stimulation at 4 Weeks (Blinded Phase)
Description: Gastrocnemius muscle endurance in response to 5 minutes of electrical stimulation therapy will be assessed with surface electromyography using a validated non-invasive device (Delsys Trino Wireless EMG System, MA, US).
Time Frame: at 4 weeks
Population: Blinded phase of study
Measure: Mean (Standard Deviation); unit: Hertz
Units Other Than Participants: lower extremities
Arm/Group | Intervention Group at 4 Weeks (Blinded Phase) | Placebo Group at 4 Weeks (Blinded Phase)
Number analyzed (Participants) | 6 | 9
Number analyzed (lower extremities) | 12 | 18
Hertz | 150.93 (7.44) | 154.44 (8.07)

12. Other Pre Specified Outcome: Frailty at 4 Weeks (Blinded Phase)
Description: Frailty will be measured with a upper-extremity wearable sensor (Frailty meter, BioSensics, MA) which enables a frailty index score based on a validated algorithm. Patients with frailty index >0.27 is considered are considered as frail. Patients with a frailty index <0.27 are considered as non-frail. The higher the frailty index, the higher the level of frailty. The frailty index ranges from 0-1.
Time Frame: up to 4 weeks
Population: blinded phase of study
Measure: Mean (Standard Deviation); unit: frailty index
Arm/Group | Intervention Group at 4 Weeks (Blinded Phase) | Placebo Group at 4 Weeks (Blinded Phase)
Number analyzed (Participants) | 11 | 13
frailty index | 0.18 (0.04) | 0.21 (0.05)

13. Other Pre Specified Outcome: Sural Nerve Conduction Velocity at 4 Weeks (Blinded Phase)
Description: Sural nerve conduction will be assessed with a DPN Check device (Neurometrix Inc, MA). The device elicits a electrical stimulation upon contact with the skin on the ankle area and returns values that can range from a minimum of 20 m/s to a maximum of 60m/s. Measurements will be obtained at 4 weeks and value will be compared between groups.
Time Frame: 4 weeks
Population: Sural nerve conduction velocity from both right and left lower extremities were measured in each participant
Measure: Mean (Standard Deviation); unit: m/s
Units Other Than Participants: lower extremities
Arm/Group | Active Group (AG) | Placebo Group (PG)
Number analyzed (Participants) | 12 | 13
Number analyzed (lower extremities) | 24 | 26
m/s | 54.96 (1.16) | 55.96 (1.40)

14. Other Pre Specified Outcome: Ankle Strength at 4 Weeks (Blinded Phase)
Description: Ankle strength will be assessed with an ankle dynamometer. Participants will be asked to perform 3 maximum voluntary contractions (MVC) sustaining ankle dorsiflexion for 5 seconds with 30 seconds of resting in between MVCs. The average of the 3 MVCs will then be calculated per lower extremity.
Time Frame: up to 4 weeks
Population: bilateral ankle strength was measured in each participant
Measure: Mean (Standard Deviation); unit: kg
Units Other Than Participants: lower extremities
Arm/Group | Active Group (AG) | Placebo Group (PG)
Number analyzed (Participants) | 12 | 13
Number analyzed (lower extremities) | 24 | 26
kg | 7.78 (0.82) | 7.93 (1.09)

15. Other Pre Specified Outcome: Plantar Tissue Oxygen Saturation at 4 Weeks (Blinded Phase)
Description: Percentage of tissue oxygen saturation (SatO2) will be measured using a validated near-infrared (NIR) camera (Snapshot NIR, KENT Imaging Inc., Calgary, AB, Can) that detects an approximate value of real-time SatO2 level in superficial tissue. The metatarsus area including the five toes will be traced.
Time Frame: up to 4 weeks
Population: blinded phase of study
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Units Other Than Participants: lower extremities
Arm/Group | Active Group (AG) | Placebo Group (PG)
Number analyzed (Participants) | 12 | 13
Number analyzed (lower extremities) | 24 | 26
percentage of oxygen saturation | 67.46 (.78) | 66.31 (.62)

16. Other Pre Specified Outcome: Mean Daily Step Count at 4 Weeks (Blinded Phase)
Description: Step count obtained with the mean 90 percentile will be will be measured over the course of the 4 weeks using a smart watch (Vivosmart 4, Garmin, US)
Time Frame: up to 4 weeks
Measure: Mean (Standard Deviation); unit: steps/day
Arm/Group | Active Group (AG) | Placebo Group (PG)
Number analyzed (Participants) | 10 | 11
steps/day | 4988.11 (3396.20) | 4887.59 (3594.30)

17. Other Pre Specified Outcome: Sleep Duration at 4 Weeks (Blinded Phase)
Description: Daily sleep duration in hours obtained with the mean 90 percentile will be measured over the course of the 4 weeks using a smart watch (Vivosmart 4, Garmin, US)
Time Frame: up to 4 weeks
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Active Group (AG) | Placebo Group (PG)
Number analyzed (Participants) | 10 | 10
hours/day | 9.2 (1.39) | 9.3 (1.2)

18. Other Pre Specified Outcome: Sural Nerve Amplitude at 4 Weeks (Blinded Phase)
Description: Sural nerve amplitude will be assessed with a DPN Check device (Neurometrix Inc, MA). The device elicits a electrical stimulation upon contact with the skin on the ankle area and returns values that can range from a minimum of 0 microVolts to a maximum of 32 microVolts. Measurements will be obtained at 4 weeks.
Time Frame: at 4 weeks
Population: Sural nerve amplitude will be measured in each of the participant's legs
Measure: Mean (Standard Deviation); unit: microVolts
Units Other Than Participants: lower extremities
Arm/Group | Intervention Group at 4 Weeks (Blinded Phase) | Placebo Group at 4 Weeks (Blinded Phase)
Number analyzed (Participants) | 10 | 12
Number analyzed (lower extremities) | 20 | 24
microVolts | 14.4 (6.23) | 16.04 (12.1)

19. Other Pre Specified Outcome: Mean Change in Functional Interference From Pain at 8 Weeks (Unblinded Phase)
Description: Pain will be assessed with a validated questionnaire called Brief Pain Inventory interference composite score (BPI-I). The maximum score is 10, meaning pain completely interferes, while the minimum score is zero, meaning pain does not interfere. This outcome assesses the difference between the mean BPI interference composite score at week 8 and week 4.
Time Frame: from week 4 to week 8
Population: week 4 to week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Intervention Group at 8 Weeks (Unblinded Phase): After 4 weeks, the IG will be unblinded, and will continue to receive high-dose TENS with a functional device for additional 4 weeks until completing 8 weeks.
  The functional device elicits 1 hour of TENS per session. Each session lasts 1 hour (100% of dose). To deliver TENS, a band strap with hydrogel pads will be placed around the calf muscle of one lower-extremity alternating to the other side in a weekly basis.
  TENS - high-dose: Subjects will receive a functional TENS device (delivers 100% of the dose) to wear for 3-5 hours per day.
- Placebo Group at 8 Weeks (Unblinded Phase): After 4 weeks, the PG will be unblinded and will switch to a high-dose TENS with a functional device for additional 4 weeks until completing 8 weeks.
  The functional device elicits 1 hour of TENS per session. Each session lasts 1 hour (100% of dose). To deliver TENS, a band strap with hydrogel pads will be placed around the calf muscle of one lower-extremity alternating to the other side in a weekly basis.
  TENS - high-dose: Subjects will receive a functional TENS device (delivers 100% of the dose) to wear for 3-5 hours per day.
Arm/Group | Intervention Group at 8 Weeks (Unblinded Phase) | Placebo Group at 8 Weeks (Unblinded Phase)
Number analyzed (Participants) | 10 | 10
score on a scale | 0.29 (2.03) | -0.87 (1.27)

20. Other Pre Specified Outcome: Mean Change in Pain Severity From 4 Weeks to 8 Weeks (Unblinded Phase)
Description: Pain severity will be assessed using the Brief Pain Inventory questionnaire composite score for severity. The maximum score is 10, meaning pain as bad as one can imagine, while the minimum score is zero, meaning no pain. This outcome assesses the difference between the mean BPI severity composite score at week 8 and week 4.
Time Frame: 4 weeks to 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group at 8 Weeks (Unblinded Phase) | Placebo Group at 8 Weeks (Unblinded Phase)
Number analyzed (Participants) | 10 | 11
score on a scale | 0.53 (1.09) | -0.43 (1.24)

21. Other Pre Specified Outcome: Mean Change in Functional Interference From Fatigue From 4 Weeks to 8 Weeks (Unblinded Phase)
Description: Functional interference from fatigue will be assessed calculating the Global Fatigue Index (GFI) obtained from a validated questionnaire called Multidimensional Assessment Fatigue, which has a minimum score of 0 (no fatigue) and a maximum sore of 100 (severe fatigue). This outcome assesses the difference between the mean global fatigue index at week 8 and week 4.
Time Frame: 4 weeks to 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group at 8 Weeks (Unblinded Phase) | Placebo Group at 8 Weeks (Unblinded Phase)
Number analyzed (Participants) | 9 | 9
score on a scale | -0.39 (7.91) | 2.14 (5.88)

22. Other Pre Specified Outcome: Stride Time at 8 Weeks During a Simple Walking Task (Unblinded Phase)
Description: as for outcome 4
Time Frame: at 8 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Intervention Group at 8 Weeks (Unblinded Phase) | Placebo Group at 8 Weeks (Unblinded Phase)
Number analyzed (Participants) | 8 | 8
seconds | 1.15 (0.10) | 1.16 (0.10)

23. Other Pre Specified Outcome: Gastrocnemius Muscle Endurance (Muscle Sustained Contraction) in Response to Electrical Stimulation at 8 Weeks (Unblinded Phase)
Description: as for outcome 11
Time Frame: at 8 weeks
Measure: Mean (Standard Deviation); unit: Hertz
Units Other Than Participants: lower extremities
Arm/Group | Intervention Group at 8 Weeks (Unblinded Phase) | Placebo Group at 8 Weeks (Unblinded Phase)
Number analyzed (Participants) | 5 | 4
Number analyzed (lower extremities) | 10 | 8
Hertz | 148.90 (6.60) | 148.52 (6.09)

24. Other Pre Specified Outcome: Frailty at 8 Weeks (Unblinded Phase)
Description: Frailty will be measured with an upper-extremity wearable sensor (Frailty meter, BioSensics, MA) which enables a frailty index score based on a validated algorithm. Patients with frailty index >0.27 is considered are considered as frail. Patients with a frailty index <0.27 are considered as non-frail. The higher the frailty index, the higher the level of frailty. The frailty index ranges from 0-1.
Time Frame: at 8 weeks
Measure: Mean (Standard Deviation); unit: frailty index
Arm/Group | Intervention Group at 8 Weeks (Unblinded Phase) | Placebo Group at 8 Weeks (Unblinded Phase)
Number analyzed (Participants) | 10 | 10
frailty index | 0.19 (0.07) | 0.19 (0.07)

25. Other Pre Specified Outcome: Sural Nerve Conduction Velocity at 8 Weeks (Unblinded Phase)
Description: Sural nerve conduction will be assessed with a DPN Check device (Neurometrix Inc, MA). The device elicits a electrical stimulation upon contact with the skin on the ankle area and returns values that can range from a minimum of 20 m/s to a maximum of 60m/s. Measurements will be obtained at 8 weeks and value will be compared between groups.
Time Frame: at 8 weeks
Measure: Mean (Standard Deviation); unit: m/s
Units Other Than Participants: lower extremities
Arm/Group | Intervention Group at 8 Weeks (Unblinded Phase) | Placebo Group at 8 Weeks (Unblinded Phase)
Number analyzed (Participants) | 7 | 7
Number analyzed (lower extremities) | 14 | 14
m/s | 55.64 (5.02) | 56.04 (5.02)

26. Other Pre Specified Outcome: Ankle Strength at 8 Weeks (Unblinded Phase)
Description: as for outcome 14
Time Frame: at 8 weeks
Measure: Mean (Standard Deviation); unit: kg
Units Other Than Participants: lower extremities
Arm/Group | Intervention Group at 8 Weeks (Unblinded Phase) | Placebo Group at 8 Weeks (Unblinded Phase)
Number analyzed (Participants) | 10 | 10
Number analyzed (lower extremities) | 20 | 20
kg | 9.59 (5.11) | 9.79 (5.18)

27. Other Pre Specified Outcome: Plantar Tissue Oxygen Saturation at 8 Weeks (Unblinded Phase)
Description: as for outcome 15
Time Frame: at 8 weeks
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Units Other Than Participants: lower extremities
Arm/Group | Intervention Group at 8 Weeks (Unblinded Phase) | Placebo Group at 8 Weeks (Unblinded Phase)
Number analyzed (Participants) | 10 | 9
Number analyzed (lower extremities) | 20 | 18
percentage of oxygen saturation | 67.82 (3.79) | 67.38 (3.38)

28. Other Pre Specified Outcome: Mean Daily Step Count at 8 Weeks (Unblinded Phase)
Description: Step count obtained with the mean 90 percentile will be will be measured starting from 4 weeks up to 8 weeks using a smart watch (Vivosmart 4, Garmin, US)
Time Frame: Starting at 4 weeks up to 8 weeks
Measure: Mean (Standard Deviation); unit: steps/day
Arm/Group | Intervention Group at 8 Weeks (Unblinded Phase) | Placebo Group at 8 Weeks (Unblinded Phase)
Number analyzed (Participants) | 2 | 5
steps/day | 3545.86 (4569.65) | 4166.31 (3897.13)

29. Other Pre Specified Outcome: Sleep Duration at 8 Weeks (Unblinded Phase)
Description: Daily sleep duration in hours obtained with the mean 90 percentile will be measured starting from 4 weeks up to 8 weeks using a smart watch (Vivosmart 4, Garmin, US)
Time Frame: Starting at 4 weeks up to 8 weeks
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Intervention Group at 8 Weeks (Unblinded Phase) | Placebo Group at 8 Weeks (Unblinded Phase)
Number analyzed (Participants) | 2 | 3
hours/day | 2.64 (1.83) | 10.53 (2.40)

30. Other Pre Specified Outcome: Sural Nerve Amplitude at 8 Weeks (Unblinded Phase)
Description: Sural nerve amplitude will be assessed with a DPN Check device (Neurometrix Inc, MA). The device elicits a electrical stimulation upon contact with the skin on the ankle area and returns values that can range from a minimum of 0 microVolts to a maximum of 32 microVolts. Measurements will be obtained at 8 weeks.
Time Frame: up to 8 weeks
Measure: Mean (Standard Deviation); unit: microVolts
Units Other Than Participants: lower extremities
Arm/Group | Intervention Group at 8 Weeks (Unblinded Phase) | Placebo Group at 8 Weeks (Unblinded Phase)
Number analyzed (Participants) | 7 | 7
Number analyzed (lower extremities) | 14 | 14
microVolts | 14.71 (7.47) | 14.71 (6.99)

31. Other Pre Specified Outcome: Double Support Phase at 4 Weeks During a Dual Walking Task (Blinded Phase)
Description: Double Support Phase will be measured with wearable sensors (LEGSys, BioSensics, MA) during a dual walking task (participants asked to count backwards by two while walking) using normal pace for 30 ft. Double support phase is defined as percentage time when both feet are simultaneously in contact with the ground during a single stride.
Time Frame: at 4 weeks
Measure: Mean (Standard Deviation); unit: percentage time
Arm/Group | Intervention Group at 4 Weeks (Blinded Phase) | Placebo Group at 4 Weeks (Blinded Phase)
Number analyzed (Participants) | 10 | 12
percentage time | 24.45 (8.47) | 24.45 (8.81)

32. Other Pre Specified Outcome: Double Support Phase at 4 Weeks During a Fast Walking Task (Blinded Phase)
Description: Double Support Phase will be measured with wearable sensors (LEGSys, BioSensics, MA) during a fast walking task (participants asked to walk at a slightly faster pace) for 30 ft. Double support phase is defined as percentage time when both feet are simultaneously in contact with the ground during a single stride.
Time Frame: at 4 weeks
Measure: Mean (Standard Deviation); unit: percentage time
Arm/Group | Intervention Group at 4 Weeks (Blinded Phase) | Placebo Group at 4 Weeks (Blinded Phase)
Number analyzed (Participants) | 11 | 11
percentage time | 17.87 (4.63) | 17.87 (4.57)

33. Other Pre Specified Outcome: Double Support Phase at 8 Weeks During a Simple Walking Task (Unblinded Phase)
Description: as for outcome 6
Time Frame: at 8 weeks
Measure: Mean (Standard Deviation); unit: percentage time
Arm/Group | Intervention Group at 8 Weeks (Unblinded Phase) | Placebo Group at 8 Weeks (Unblinded Phase)
Number analyzed (Participants) | 8 | 8
percentage time | 20.69 (4.77) | 21.75 (4.13)

34. Other Pre Specified Outcome: Double Support Phase at 8 Weeks During a Dual Task (Unblinded Phase)
Description: as for outcome 31
Time Frame: at 8 weeks
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Intervention Group at 8 Weeks (Unblinded Phase) | Placebo Group at 8 Weeks (Unblinded Phase)
Number analyzed (Participants) | 9 | 7
percentage | 24.47 (3.24) | 24.51 (2.27)

35. Other Pre Specified Outcome: Stride Time at 8 Weeks During a Dual Task (Unblinded Phase)
Description: as for outcome 9
Time Frame: at 8 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Intervention Group at 8 Weeks (Unblinded Phase) | Placebo Group at 8 Weeks (Unblinded Phase)
Number analyzed (Participants) | 9 | 7
seconds | 1.21 (0.15) | 1.27 (0.15)

36. Other Pre Specified Outcome: Stride Time at 8 Weeks During a Fast Walk Task (Unblinded Phase)
Description: as for outcome 10
Time Frame: at 8 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Intervention Group at 8 Weeks (Unblinded Phase) | Placebo Group at 8 Weeks (Unblinded Phase)
Number analyzed (Participants) | 8 | 7
seconds | 0.99 (0.11) | 1.04 (0.10)

37. Other Pre Specified Outcome: Cadence at 8 Weeks During a Simple Walking Task (Unblinded Phase)
Description: as for outcome 5
Time Frame: at 8 weeks
Measure: Mean (Standard Deviation); unit: steps/min
Arm/Group | Intervention Group at 8 Weeks (Unblinded Phase) | Placebo Group at 8 Weeks (Unblinded Phase)
Number analyzed (Participants) | 8 | 8
steps/min | 105.36 (10.16) | 101.63 (5.77)

38. Other Pre Specified Outcome: Cadence at 8 Weeks During a Dual Task (Unblinded Phase)
Description: as for outcome 7
Time Frame: at 8 weeks
Measure: Mean (Standard Deviation); unit: steps/min
Arm/Group | Intervention Group at 8 Weeks (Unblinded Phase) | Placebo Group at 8 Weeks (Unblinded Phase)
Number analyzed (Participants) | 9 | 7
steps/min | 100.51 (12.56) | 96.04 (10.62)

39. Other Pre Specified Outcome: Cadence at 8 Weeks During a Fast Walking Task (Unblinded Phase)
Description: as for outcome 8
Time Frame: at 8 weeks
Measure: Mean (Standard Deviation); unit: steps/min
Arm/Group | Intervention Group at 8 Weeks (Unblinded Phase) | Placebo Group at 8 Weeks (Unblinded Phase)
Number analyzed (Participants) | 8 | 7
steps/min | 122.80 (14.88) | 116.14 (12.59)

ADVERSE EVENTS:
Time Frame: AEs were collected from study start date (March 1 2022) to the study completion (December 1, 2023) in a non-systematic way. Per patient, AEs were collected up to 8 weeks after Baseline. During follow-ups, participants were asked if they experienced AEs. If participant missed a visit or had low adherence (assessed by monitoring device usage remotely) the coordinator called the participant and asked for AEs. AEs were also reported by the participants on a case-by-case basis when they occurred.
Description: The clinicaltrials.gov definitions were used. We collected unfavorable medical occurrences experienced by study participants and noted whether they were study device related (caused directly by the device), unrelated to the study device, or whether it was caused by improper device usage. This information was collected non-systematically and not separately -- either participants reported events directly or during phone calls/study visits study coordinators asked about issues.
Arm/Group | Intervention Group at 4 Weeks (Blinded Phase) | Placebo Group at 4 Weeks (Blinded Phase) | Intervention Group at 8 Weeks (Unblinded Phase) | Placebo Group at 8 Weeks (Unblinded Phase)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 3/15 | 3/15 | 0/12 | 0/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Group at 4 Weeks (Blinded Phase) (N=15) | Placebo Group at 4 Weeks (Blinded Phase) (N=15) | Intervention Group at 8 Weeks (Unblinded Phase) (N=12) | Placebo Group at 8 Weeks (Unblinded Phase) (N=13)
Minor AE due to device misuse (Product Issues) | 3 | 3 | 0 | 0 — Incorrect device placement or using device for longer than instructed led to some expressing pain, fatigue, skin irritation, rash, or itchiness were experienced. These were resolved once device usage adjusted to follow instructions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/58/NCT05200858/Prot_SAP_000.pdf
  • Informed Consent Form (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/58/NCT05200858/ICF_001.pdf